CLINICAL TRIAL: NCT02102854
Title: Single Dose rATG for Treatment of Acute Renal Allograft Rejection
Brief Title: Single Dose rATG for Renal Allograft Rejection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Samir J. Patel, Clinical Pharmacist, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003442; 0809-0111 (Other: HMRI IRB)
Record Dates: First submitted 2014-03-26; First posted 2014-04-03 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Acute (Cellular) Renal Allograft Rejection
Keywords: kidney transplantation; acute rejection; rabbit antithymocyte globulin
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dose rATG (Active Comparator): Standard dose rATG given as daily infusions of 1.5 mg/kg x 4-5 days
  Interventions: Drug: rATG
- Single dose rATG (Experimental): Single dose rATG give as 2 consecutive 3 mg/kg IV infusions to be completed over a 24-36 hour duration
  Interventions: Drug: rATG

INTERVENTIONS:
Drug: rATG — Infusion of horse or rabbit-derived antibodies against human T cells, used to prevent & treat acute rejection in organ transplantation
  Other Names: Rabbit antithymocyte globulin; Thymoglobulin; ATG

SUMMARY:
Rabbit antithymocyte globulin (rATG) is approved for the treatment of acute rejection following kidney transplantation and is routinely administered as a series of 5-7 consecutive daily doses via central intravenous catheter.Single large-doses of rATG have been shown to have equivalent safety and efficacy profile compared to the standard daily protocol when used as an induction agent but there are no reported experiences of its use for rejection treatment. Plan to study a single-dose rATG infusion compared to standard rATG administration including correlation to length of hospital stay and hospital costs.

DETAILED DESCRIPTION:
Rabbit antithymocyte globulin (rATG) is approved for the treatment of acute rejection following kidney transplantation and is routinely administered as a series of 5-7 consecutive daily doses via central intravenous catheter. This prolonged course is not consistent with the Medicare diagnosis-related group (DRG) for acute rejection which limits rejection admission to 3 days. The prolonged hospitalization results in increased medical costs and uniform financial loss to the hospital for patients admitted under this DRG. In addition there is a patient related toll of the prolonged hospitalization and a potential for additional hospital acquired complications. Single large-doses of rATG have been shown to have equivalent safety and efficacy profile compared to the standard daily protocol when used as an induction agent but there are no reported experiences of its use for rejection treatment. The investigators hypothesize that single-dose rATG infusion will be as safe and efficacious as standard rATG administration when used for rejection treatment and would result in significant reduction in the length of hospital stay (LOS) and hospital costs for rejection treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older
2. Experiencing a biopsy-proven acute rejection episode which:

   * will require the use of rATG based on severity, or
   * is exhibiting resistance to corticosteroid treatment, defined as failure of the serum creatinine to decrease after at least 3 days of corticosteroid treatment (≥200 mg/day of methylprednisolone or equivalent)

Exclusion Criteria:

1. Patients with known severe allergy to antithymocyte globulin or rabbits
2. Rejection episode requiring the use of therapeutic plasma exchange immediately subsequent to rATG administration
3. Currently receiving any investigational drug or treatments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2021-03 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Hospital length of hospitalization (days) | 7 days
  The length of hospitalization for treatment of renal allograft rejection in days will be determined which should be an average of 5-7 days

SECONDARY OUTCOMES:
Infusion related symptoms | 7 days
  Incidence of grade 1, 2, or 3 infusion-related symptoms, graded according to common terminology criteria will be determined during the patient's hospital admission, which should be an average of 5-7 days

OTHER OUTCOMES:
Rate of 30-day readmissions (%) | 30 days
  Proportion of participants re-admitted to the hospital from discharge to day 30 for each group
Incidence of leukopenia | 6 months
  Incidence leukopenia, graded according the to common terminology criteria
Incidence of neutropenia (%) | 6 months
  Incidence of neutropenia, graded according the to common terminology criteria
Incidence of thrombocytopenia (%) | 6 months
  Incidence of thrombocytopenia, graded according the to common terminology criteria
Incidence of BK viremia (%) | 6 months
  Incidence of BK viremia or nephropathy at 6 months
Incidence of cytomegalovirus (CMV) viremia (%) | 6 months
  Incidence of CMV viremia or disease at 6 months
Non-hematologic adverse events (%) | 6 months
  Non-hematologic adverse events (i.e. serum sickness)
Clinical reversal of rejection | 6 months
  Clinical reversal of rejection, defined as the return of serum creatinine to pre-rejection creatinine
Time to reversal of rejection | 6 months
  Number of days to reversal of rejection
Histological reversal of rejection | 6 months
  Biopsy demonstrated absence of rejection if available
Kidney function status at 1, 3 and 6 months post-rejection treatment | 6 months
  Serum creatinine at 1, 3 and 6 months post-rejection treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samir Patel, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No